CLINICAL TRIAL: NCT06036264
Title: Monocentric Retrospective Cohort Study of the Impact of Advanced Nursing Practice on the Follow-up of the End Stage Chronic Renal Disease Patient: Influence on the Implementation of an Arteriovenous Fistula Prior to Dialysis and on Access to Renal Transplantation
Brief Title: Monocentric Retrospective Cohort Study of the Impact of Advanced Nursing Practice on the Follow-up of the End Stage Chronic Renal Disease Patient
Acronym: IPASIRC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN132022/CHUSTE
Record Dates: First submitted 2023-08-21; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-02

CONDITIONS: Renal Disease
Keywords: advanced practice nurse; kidney transplantation; renal disease; arteriovenous fistula; Chronic Kidney Disease
MeSH Terms: conditions — Kidney Diseases; Arteriovenous Fistula; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Exposed subject group: Patients, starting dialysis, eligible for arteriovenous fistula (AVF) creation and/or renal transplantation who received pre-Advanced Practice Nurse (APN) intervention in their care pathway will be included Datas will be collected of medical record.
  Interventions: Other: Collected of Datas
- Comparable unexposed subject group: All patients starting dialysis sessions eligible for arteriovenous fistula (AVF) creation and/or renal transplantation will be included.
  Datas will be collected of medical record.
  Interventions: Other: Collected of Datas
- professional working with the pre-Advanced Practice Nurse (APN): professional working with the pre-Advanced Practice Nurse (APN) will be included.
  Semi-structured interview will be performed.
  Interventions: Other: semi-structured interview

INTERVENTIONS:
Other: Collected of Datas — age, sex, mode of dialysis, emergency context, approach, date of creation of the arteriovenous fistula (if concerned), date of start of dialysis, transplant status, date of registration on the renal transplant waiting list (if concerned), nephrologist, date of first consultation with the pre-nurse in advanced practice (APN) (if concerned)
  Groups: Comparable unexposed subject group; Exposed subject group
Other: semi-structured interview — Semi-structured interviews will be realized. The goal is to establish a qualitative analysis of the relevance and organization of pre-transplant assessments, of the reactivity in the adjustment of requests and assessments, and to identify the strong points or areas for improvement.
  Groups: professional working with the pre-Advanced Practice Nurse (APN)

SUMMARY:
With regard to the fields of competence of advanced practice defined by the Order of October 22, 2021 amending the Order of July 18, 2018 on the system of studies for the State diploma of advanced practice nurse mentioning renal disease, dialysis and renal transplantation (MRDT) and the latest recommendations of the French National Authority for Health (HAS) of July 1 2021 on the monitoring of patients with Chronic Kidney Disease (CKD), the Advanced Practice Nurse (APN) has its place in improving practices and the care pathway of patients suffering from end-stage chronic renal failure (CKD).

In the literature, there are a number of studies arguing the benefits of advanced practice nurse follow-up with patients suffering from chronic renal failure (CKD) in terms of improving their psycho-social and self-care skills. However, few studies, particularly in France, demonstrate its role in the coordination of care. By virtue of their training, advanced practice nurse with an disease, dialysis and renal transplantation (MRDT) specialization acquire skills in managing pretransplant assessment files and in planning the creation of arteriovenous fistula (AVF), which enable them to be autonomous and relevant professionals in the coordination of these processes. This is why it seems appropriate to look at the added value that advanced nursing practice can bring to the follow-up of these patients.

DETAILED DESCRIPTION:
To this end, a study of the practices and social representations of healthcare professionals involved in the management of Chronic Kidney Disease (CKD) patients can allow us to - To explore current practices under the focus of follow-up by a nephrologist and an advanced nurse on access to renal transplantation and on the implementation of arteriovenous fistula (AVF) versus follow-up by a nephrologist only.

* To perceive the "reading grids" that health professionals in transplant centers assign to the management of this type of patient by an Advanced Practice Nurse (APN).
* To question the identity issues associated with the actors by taking into account their status and roles in the institution and in interdisciplinaritý.

This study should produce initial results on the changes induced by advanced nursing practice on access to care and on the improvement of complex care pathways and more particularly for the Chronic Kidney Disease (CKD) patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients starting dialysis sessions
* Patient eligible for arteriovenous fistula (AVF) and/or renal transplantation who started dialysis sessions between January 1st 2016 and December 31st 2021 at the Roanne Hospital.

Exclusion Criteria:

* Patient starting dialysis in emergency without prior nephrological followup.
* Patients who started dialysis in other dialysis centers (transfer: no knowledge of their previous nephrological follow-up)
* Patients starting dialysis at dates earlier or later than those determined in the study.
* Patients with missing data at the time of data collection.
* Patients under legal protection (guardianship, curatorship) or with cognitive impairment preventing informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient eligible for arteriovenous fistula (AVF) and/or renal transplantation who started dialysis sessions between January 1st 2016 and December 31st 2021 at the Roanne Hospital will be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the impact of the implementation of an Advanced Practice Nurse (APN) dedicated to the nephrology care pathway on the creation of arteriovenous fistula before dialysis sessions. | Year: 1
  Rate of patients arriving with a functional arteriovenous fistula (AVF) at dialysis start. This rate will be compared between patients starting dialysis who received alternating nephrologist/pre-Advanced Practice Nurse (APN) follow-up and patients starting dialysis who received usual follow-up (control group).

SECONDARY OUTCOMES:
Rate of patients on the transplant list. | Year: 1
  This rate will be compared between patients starting dialysis who received alternating nephrologist/pre-IP follow-up and patients starting dialysis who received usual follow-up (control group).
To explore the beliefs and attitudes of healthcare professionals in transplant centers regarding the management of patients by an Advanced Practice Nurse (APN). | Year: 1
  Analysis semi-structured interviews results.
Identify the strengths and areas for improvement of this system. | Year: 1
  Analysis semi-structured interviews results.
Rate of patients on the transplant list | Year: 1
  This rate will be compared between patients starting dialysis who received alternating nephrologist/pre-Advanced Practice Nurse (APN) follow-up and patients starting dialysis who received usual follow-up (control group).
To explore the "reading grids" that healthcare professionals in transplant centers assign to the intervention of the Advanced Practice Nurse (APN) in the management of chronic renal failure (CKD) patients. | Year: 1
  Analysis semi-structured interviews results.
Isolate the obstacles and facilitators to the intervention of Advanced Practice Nurse (APN) in this care pathway | Year: 1
  Analysis semi-structured interviews results.

CONTACTS AND LOCATIONS:
Overall Officials: Françoise RAY, Nurse, Principal Investigator — Centre Hospitalier de Roanne
Locations (1):
- CH de Roanne, Roanne, France

IPD SHARING:
Plan to Share IPD: No